CLINICAL TRIAL: NCT00411060
Title: Orthopaedic Data Bank; Collection and Storage of Data Relating to Orthopaedic Disorders
Brief Title: Clinical Orthopaedic Data Bank (Acute and Chronic)
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201501013; 117-2006 (Other: Legacy study); OCR18422 (Other: Universiy of Florida)
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis; Osteosarcoma; Scoliosis; Cerebral Palsy
Keywords: Rotator Cuff Tear
MeSH Terms: conditions — Osteoarthritis; Osteosarcoma; Scoliosis; Cerebral Palsy; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data involving orthopaedic conditions and rehabilitation aspects of musculoskeletal and neuromuscular disorders will be collected and stored as part of the normal clinical care of patients seen in the University of Florida (UF) and Shands Orthopaedics and Sports Medicine Institute.

DETAILED DESCRIPTION:
All patients seen the Orthopaedic clinic will be informed of the data collection and asked to participate. If the patient is agreeable to participation, informed consent will then be obtained.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen in the UF&Shands Orthopaedics and Sports Medicine Institute will be asked to sign an informed consent.

Exclusion Criteria:

* No exclusions, all patients interested in participation will be asked to sign an informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Orthopaedic clinic
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2007-01; Primary Completion 2026-08-14 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Retrospective data | 2007 to present, until 2020
  Medical Record information will be used as needed for a future IRB retrospective study

CONTACTS AND LOCATIONS:
Overall Officials: Parker Gibbs, MD, Principal Investigator — UF Department of Orthopaedics and Rehabilitation
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

REFERENCES:
- See also: University of Florida Department of Orthopaedics Research — http://www.ortho.ufl.edu